CLINICAL TRIAL: NCT04744506
Title: Targeted Axillary Dissection Using Carbon Marking for Patients With Node-positive Breast Cancer Following Neoadjuvant Therapy (TADCOM): a Prospective, Multicenter, Randomized Controlled Trial
Brief Title: Targeted Resection of Axillary Metastatic Lymph Nodes After Breast Cancer Neoadjuvant Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Provincial Natural Science Foundation of China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-535
Record Dates: First submitted 2020-12-27; First posted 2021-02-09 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer; Surgery; Lymph Node Metastases
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Intervention Model Description: Group 1: CG-TAD Group (Control) US-guided clip insertion into suspicious ALNs pre-NAC Post-NAC, TAD removing SLNs and clipped LNs Group 2: CN-LNM Group US-guided CNSI injection to tattoo suspicious ALNs pre-NAC Post-NAC, TAD removing SLNs and carbon-marked LNs Group 3: PCN-MAP Group US-guided CNSI injection around primary tumor pre-NAC, additional US-guided clip placement for metastatic LN Post-NAC, TAD removing SLNs, carbon-marked LNs, and clipped LNs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: CG-TAD Group (Active Comparator): US-guided clip insertion into suspicious ALNs pre-NAC Post-NAC, TAD removing SLNs and clipped LNs
  Interventions: Device: Tissue Marker Clip
- Group 2: CN-LNM Group (Experimental): US-guided CNSI injection to tattoo suspicious ALNs pre-NAC Post-NAC, TAD removing SLNs and carbon-marked LNs
  Interventions: Drug: Carbon Nanoparticle Suspension Injection
- Group 3: PCN-MAP Group (Experimental): US-guided CNSI injection around primary tumor pre-NAC, additional US-guided clip placement for metastatic LN Post-NAC, TAD removing SLNs, carbon-marked LNs, and clipped LNs
  Interventions: Drug: Carbon Nanoparticle Suspension Injection

INTERVENTIONS:
Device: Tissue Marker Clip — Tissue Marker Clip to be Placed in Metastatic Axillary Lymph Node (Before Neoadjuvant Chemotherapy for Breast Cancer)
  Arms: Group 1: CG-TAD Group
Drug: Carbon Nanoparticle Suspension Injection — Carbon Nanoparticle Suspension Injection to be Placed in Metastatic Axillary Lymph Node (Before Neoadjuvant Chemotherapy for Breast Cancer)
  Arms: Group 2: CN-LNM Group
Drug: Carbon Nanoparticle Suspension Injection — Carbon Nanoparticle Suspension Injection to be Placed around Primary Tumor (Before Neoadjuvant Chemotherapy for Breast Cancer)
  Arms: Group 3: PCN-MAP Group

SUMMARY:
This study evaluates the efficacy and feasibility of Carbon Nanoparticle Suspension Injection (CNSI) for Targeted Axillary Dissection (TAD) in breast cancer patients undergoing neoadjuvant chemotherapy (NAC), compared to traditional clip-based methods. By leveraging CNSI's enhanced visibility and stability, the study aims to improve the precision of lymph node removal, reduce surgical complications, and potentially transform clinical practices. Conducted across multiple centers, this randomized controlled trial focuses on clinical outcomes such as lymph node retrieval rates and the accuracy of surgical staging, aiming to establish a safer, more effective approach to managing axillary lymph nodes in breast cancer surgery.

DETAILED DESCRIPTION:
Objective: This study aims to assess the clinical feasibility, accuracy, and effectiveness of CNSI in targeted axillary dissection compared to traditional tissue marker clips in patients with breast cancer undergoing neoadjuvant chemotherapy (NAC).

Background: Breast cancer remains one of the most prevalent cancers among women globally. Neoadjuvant chemotherapy (NAC) has significantly advanced the management of locally advanced breast cancer, enabling more conservative surgical approaches and reducing the dependency on axillary lymph node dissection (ALND), which is often associated with long-term complications such as lymphedema and chronic pain. Traditional TAD methods using tissue marker clips have challenges including high costs and potential for marker loss. CNSI presents a novel approach with potential for enhanced surgical precision and reduced complication rates.

Methods: The study employs a multicenter, randomized controlled trial design to compare the outcomes of TAD using CNSI versus conventional clip-based methods. Patients with clinically node-positive breast cancer who achieve clinical node-negative status post-NAC are enrolled. The primary endpoints include the rate of successful lymph node retrieval, the incidence of surgical complications, and the accuracy of lymph node staging.

Innovation: CNSI is designed to improve the visibility and stability of lymph nodes during surgery, potentially increasing the precision of cancerous node removal and minimizing the need for subsequent surgical interventions. Its unique properties, such as the slow metabolic rate and strong pigmentation, ensure prolonged visibility and facilitate easier identification during surgery.

Significance: By enhancing the effectiveness of TAD, CNSI could transform clinical practices in breast cancer surgery, reducing the physical burden of surgery and improving the quality of life for patients. The study's findings could lead to broader adoption of CNSI in surgical oncology, setting a new standard for axillary management in breast cancer.

Conclusion: This research could significantly impact breast cancer treatment protocols by providing a safer, more cost-effective, and clinically advantageous method for axillary lymph node management, potentially leading to widespread changes in surgical approaches and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18 to 85 years are eligible.
2. Participants must have a histologically confirmed diagnosis of breast cancer, classified as cT1-4N1-2aM0 according to the 8th edition of the AJCC (American Joint Committee on Cancer) TNM classification system.
3. Eastern Cooperative Oncology Group (ECOG) performance status must be 0 or 1.
4. Clinical re-staging must indicate an axillary node status of ycN0 following NAC.
5. Participants must provide written informed consent to partake in the trial, acknowledging understanding and agreement to the procedures and risks involved.

Exclusion Criteria:

1. Patients with metastatic breast cancer (Stage IV).
2. Diagnosed with inflammatory breast cancer or bilateral breast cancer.
3. History of axillary surgical procedures.
4. Any medical, psychological, or social conditions that would prevent adherence to the study protocol or completion of the treatment or follow-up.
5. Known allergy to carbon nanoparticles or presence of severe comorbid conditions or other serious underlying medical issues.
6. Current or prior participation in another clinical trial that could interfere with the outcome of this study or affect the safety and well-being of the participants.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2028-07-15 (Estimated); Study Completion 2029-07-15 (Estimated)

PRIMARY OUTCOMES:
Lymph node retrieval rate marked | Up to 2 months
  The proportion of successfully retrieved marked lymph nodes will be calculated and compared among the study groups to evaluate the effectiveness of each marking technique.
Number of sentinel and marked lymph nodes | Up to 2 months
  The mean, median, and range of the number of sentinel and marked lymph nodes harvested during surgery will be recorded and compared to assess the efficacy of the marking techniques in identifying lymph nodes of interest.
Concordance between marked and sentinel lymph nodes | Up to 2 months
  The consistency between marked lymph nodes and intraoperatively identified sentinel lymph nodes will be evaluated by calculating the percentage of marked nodes that are also sentinel nodes and vice versa.
Complication rate | Up to 60 months
  All surgery-related complications, including but not limited to hemorrhage, lymphedema, infection, pain, tissue damage, clip displacement, clip loss, absence of CNSI staining, and excessive CNSI staining, will be recorded and analyzed. The overall complication rate and rates for specific types of complications will be reported. The severity of complications will be assessed using the Clavien-Dindo classification to provide a standardized evaluation of complication severity.

SECONDARY OUTCOMES:
Axillary and distant recurrence rates | Up to 60 months
  During the 2-year and 5-year follow-up periods, the axillary and distant recurrence rates will be monitored and reported for each study group to assess the long-term oncological outcomes of the different marking techniques.
Overall survival (OS), and disease-free survival (DFS) | Up to 60 months
  OS and DFS will be monitored and reported for each study group at 2 years, 5 years, and other relevant time points. Kaplan-Meier analysis and Cox proportional hazards models will be used to estimate these endpoints and compare outcomes among the study groups.
Surgical duration | Up to 2 hours
  The total time from the start of the surgery to the removal of the last lymph node will be calculated to analyze the efficiency of different techniques in terms of surgical time.
Postoperative complications | Up to 60 months
  Complications such as lymphedema, infection, and pain will be assessed at specific time points (e.g., 1 month, 6 months, and 1 year post-surgery) using validated tools or scales (e.g., Common Terminology Criteria for Adverse Events, Brief Pain Inventory) to determine the safety profile of each marking technique and its impact on patient morbidity.
The Life Quality Index | Up to 24 months
  The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Breast Cancer Module 23 (EORTC QLQ-BR23) will be used to evaluate patients' quality of life before treatment, at 6 months, 1 year, and 2 years after treatment to assess the impact of the different marking techniques on patient-reported outcomes.
Positive tumor margin rate and re-excision surgery | Up to 6 months
  For patients undergoing breast-conserving surgery, the proportion of positive tumor margins, defined as tumor cells at the inked margin or within 1 mm from the margin, will be evaluated postoperatively. The rate of re-excision surgery due to positive margins will also be assessed to evaluate the impact of the marking techniques on the accuracy of surgical resection and the need for additional interventions.

CONTACTS AND LOCATIONS:
Overall Officials: Huang Jian, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen W, Pang L, Jin X, Chen H, Huang J. Targeted axillary dissection using carbon marking for patients with node-positive breast cancer following neoadjuvant therapy (TADCOM): study protocol for a prospective, multicenter, randomized controlled trial. BMC Cancer. 2024 Oct 15;24(1):1276. doi: 10.1186/s12885-024-13001-2. PMID 39402559

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04744506/Prot_SAP_002.pdf
  • Informed Consent Form (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/06/NCT04744506/ICF_003.pdf